CLINICAL TRIAL: NCT03515850
Title: Clinical Trial of Anatomical Classifications of Inferior Mesenteric Artery in Laparoscopic Rectal Resection Surgery
Brief Title: Anatomical Classifications of Inferior Mesenteric Artery
Acronym: IMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Li Chuan (Other)
Responsible Party: Sponsor-Investigator, Li Chuan, Southwest Hospital, China, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Other Study IDs: Southwest-IMA-rectal
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2018-05-04 (Actual); Status verified 2018-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The vascular branches of inferior mesenteric artery (IMA) involve superior rectal artery(SRA),Sigmoid artery(SA) and the left colic artery(LCA). Different levels of ligation of the (IMA) are applied in rectal cancer surgery, including retain or not retain the left colic artery(LCA). Retained the LCA would facilitate the vascularity. The variations of vessels are more frequent in the combinations of branches, while LCA, SA and SRA may vary from people to people. Which contribute to the difficulty of surgery to retain the LCA.. As a result, a better understanding of the anatomical branches classification of IMA is a must during operation. However, existing studies of IMA's branches combination are very rare and often single-centered with minimal samples. In order to achieve better surgical outcome and reduce operative complications, the investigators design this study to investigate the anatomical classification of IMA and the surgical outcome of each type

ELIGIBILITY:
Inclusion Criteria:

1. Patients who undergoing laparoscopic rectal cancer surgery.
2. Pathology: adenocarcinoma or huge adenomas proven by colonoscopic biopsy.
3. Localization: tumor located between distal sigmoid colon and anal canal.
4. Patients have to be aware of the aim of the trial, and have signed the informed consent.

Exclusion Criteria:

1. History of any gastrointestinal surgery.
2. Patients with emergent surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective study，and based on the conjoin classifications of branches, the anticipant populations of this study is 500.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-05 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
classifications vascular branches of IMA | 3years
  based on the positon of LCA that conjoin the IMA

CONTACTS AND LOCATIONS:
Locations (1):
- General Surgery Center of PLA, Chongqing, China